CLINICAL TRIAL: NCT01535235
Title: ACE Inhibitors to Decrease Lymphoid Fibrosis in Antiretroviral-Treated, HIV-infected Patients: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-08132
Record Dates: First submitted 2012-02-09; First posted 2012-02-17 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: HIV
Keywords: HIV; Lymphoid fibrosis
MeSH Terms: interventions — Lisinopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACE Inhibitor (Active Comparator): Active group
  Interventions: Drug: Lisinopril
- Placebo (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisinopril — Lisinopril 20mg QD x 24 weeks
  Arms: ACE Inhibitor
Drug: Placebo — Placebo QD x24wks
  Arms: Placebo

SUMMARY:
The investigators propose a proof-of-concept, pathogenesis-oriented, randomized, placebo-controlled pilot study to assess whether the addition of an angiotensin converting enzyme (ACE) inhibitor to standard Highly Active Antiretroviral Therapy (HAART) reverses lymphoid fibrosis, and whether this leads to more effective HIV-specific host immune responses and an accelerated clearance of the latent reservoir.

ELIGIBILITY:
Inclusion Criteria include:

* Stable HAART with maintenance of plasma HIV RNA levels below level of detection (< 40-75 copies/mL) for ≥ 12 months
* > 90% adherence to HAART within preceding 30 days

Exclusion Criteria include:

* Screening systolic blood pressure < 110mm Hg or diastolic blood pressure < 60mm Hg
* Current use of any ACE inhibitor, angiotensin receptor blocker, or aldosterone antagonist
* Known diabetes mellitus or cardiovascular/kidney/collagen vascular disease
* Pregnant/breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyu Hatano, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial over enrolled by one individual as one participant discontinued the study after enrollment due to an adverse event.
Period: Overall Study
Arm/Group | ACE Inhibitor | Placebo
Started | 16 | 15
Completed | 15 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- ACE Inhibitor: Active group
  Lisinopril: Lisinopril 20mg Daily x 24 weeks
- Placebo: Placebo group
  Placebo: Placebo Daily x24wks
- Total: Total of all reporting groups
Arm/Group | ACE Inhibitor | Placebo | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [45.5 to 56] | 54 [47 to 58] | 54 [47 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 15 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  White | 14 | 9 | 23
  Black/African American | 2 | 1 | 3
  Hispanic/Latino | 0 | 3 | 3
  Asian | 0 | 1 | 1
  Pacific Islander | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31
CD4+ T cell count [Median (Inter-Quartile Range); unit: cells/mm^3] | 349 [230 to 415] | 392 [237 to 641] | 362 [237 to 636]

OUTCOME MEASURES:

1. Primary Outcome: Change in HIV RNA (Copies/Million Rectal Cells)
Description: Change in HIV RNA measured in GALT (gut-associated lymphoid tissue) from baseline
Time Frame: 22 weeks
Population: Three participants in the placebo group did not have sufficient cells for analysis for one of the time points.
Measure: Median (Inter-Quartile Range); unit: copies/million rectal cells
Arm/Group | ACE Inhibitor | Placebo
Number analyzed (Participants) | 15 | 12
copies/million rectal cells | 1.1 [-74.5 to 62.5] | -0.2 [-55.8 to 96.4]
Statistical Analysis 1: Comparison: ACE Inhibitor vs Placebo; Test type: Superiority or Other; p = 0.63, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in HIV DNA (Copies/Million Rectal Cells)
Description: Change in HIV DNA measured in GALT (gut-associated lymphoid tissue) from baseline
Time Frame: 22 weeks
Population: Three participants in the placebo group did not have sufficient cells for analysis for one of the time points.
Measure: Median (Inter-Quartile Range); unit: copies/million rectal cells
Arm/Group | ACE Inhibitor | Placebo
Number analyzed (Participants) | 15 | 12
copies/million rectal cells | -38.4 [-76.3 to 114.8] | -53.8 [-102.9 to 87.3]
Statistical Analysis 1: Comparison: ACE Inhibitor vs Placebo; Test type: Superiority or Other; p = 0.63, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | ACE Inhibitor | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 1/16 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACE Inhibitor (N=16) | Placebo (N=15)
Elevation in serum creatinine (Renal and urinary disorders) | 1 (1) | 0 (0) — One subject had elevation of serum creatinine and was withdrawn from the study at Week 12 for this. However, labs drawn at that time showed that the serum creatinine had returned to baseline and was likely secondary to another medical condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No